CLINICAL TRIAL: NCT00149747
Title: Promoting Exercise, Sleep and Well-Being in Older Adults
Brief Title: The Effectiveness of Regular Exercise on Improving Sleep in Older Adults
Acronym: RTC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Abby C King, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH058853 (NIH); R01MH058853 (NIH); DAHBR HB-C
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Initiation and Maintenance Disorders; Sleep Disorders, Intrinsic
Keywords: Sleep; Exercise; Older Adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Intrinsic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training (Experimental): Group based exercise training. Two weekly classes including aerobic endurance physical activity and strength and flexibility training, and up to three home-based sessions of similar composition of aerobic endurance, strength and flexibility training.
  Interventions: Behavioral: Moderate-Intensity Aerobic Physical Activity
- 2 (Placebo Comparator): Attention-control of exposure to study staff. Weekly general health education classes conducted in group sessions.
  Interventions: Behavioral: Health Education Class

INTERVENTIONS:
Behavioral: Moderate-Intensity Aerobic Physical Activity — Moderate-Intensity Aerobic Physical Activity. 4+ days per week, 60+ minutes per day, moderate or greater intensity physical activity
  Other Names: Comprehensive fitness class
  Arms: Exercise training
Behavioral: Health Education Class — 2 classes a week, 90+minutes per class, general health education, excluding information on physical activity
  Other Names: Healthy Aging Workshops
  Arms: 2

SUMMARY:
This study will evaluate the effect of regular aerobic exercise on improving sleep in older adults with moderate difficulty sleeping.

DETAILED DESCRIPTION:
Sleep deprivation is a common problem among older adults. It is often at the root of increased mortality and some psychiatric disorders. Regular participation in a medium-intensity exercise regimen may help people sleep better. This study will assess the effectiveness of a regular exercise program on improving sleep in older adults with moderate difficulty sleeping.

Participants will be randomly assigned to one of two conditions. One group will partake in a moderate-intensity physical activity training regimen. The other group will act as a non-exercise attention-control comparison group. Each group will undergo its assigned treatment for 12 months. Sleep quantity and quality will be measured objectively using in-home polysomnography. Subjective sleep quality and health-related quality of life measures will be evaluated with questionnaires. All measurements will be performed at the beginning of the study, Month 6, and Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Moderate difficulty sleeping unrelated to a physical illness or psychopathology (determined by the Sleep Questionnaire and Assessment of Wakefulness)
* Currently not physically active on a regular basis
* Body mass index less than 38

Exclusion Criteria:

* Currently physically active on a regular basis
* Diagnosed with a clinically significant sleep disorder
* Mild or no sleep complaints (determined by the Sleep Questionnaire and Assessment of Wakefulness)
* Unstable on medications
* Current smoker
* Consumes more than three alcoholic beverages per day
* Medical condition that may limit participation in moderate-intensity exercise
* Diagnosed with clinical psychopathology

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 1999-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby C King, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Prevention Research Center, Stanford, California, United States

REFERENCES:
- [Background] King AC, Oman RF, Brassington GS, Bliwise DL, Haskell WL. Moderate-intensity exercise and self-rated quality of sleep in older adults. A randomized controlled trial. JAMA. 1997 Jan 1;277(1):32-7. PMID 8980207
- [Background] Bliwise DL, King AC, Harris RB, Haskell WL. Prevalence of self-reported poor sleep in a healthy population aged 50-65. Soc Sci Med. 1992 Jan;34(1):49-55. doi: 10.1016/0277-9536(92)90066-y. PMID 1738856
- [Result] King AC, Pruitt LA, Woo S, Castro CM, Ahn DK, Vitiello MV, Woodward SH, Bliwise DL. Effects of moderate-intensity exercise on polysomnographic and subjective sleep quality in older adults with mild to moderate sleep complaints. J Gerontol A Biol Sci Med Sci. 2008 Sep;63(9):997-1004. doi: 10.1093/gerona/63.9.997. PMID 18840807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited through radio and newspaper advertisement, direct mailings to local addresses.
Pre-assignment Details: Overnight pulse oximetry for 1 night to rule out sleep apnea
Groups:
- Exercise Group: Regular, aerobic endurance physical activity
  Moderate-Intensity Aerobic Physical Activity : 4+ days per week, 60+ minutes per day, moderate or greater intensity physical activity
- Attention-Control (Health Education) Group: Weekly general health education classes
  Health Education Class : 2 classes a week, 90+minutes per class, general health education, excluding information on physical activity
Period: Overall Study
Arm/Group | Exercise Group | Attention-Control (Health Education) Group
Started | 36 | 30
Completed | 32 | 27
Not Completed | 4 | 3
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Attention-Control (Health Education) Group | Total
Number analyzed (Participants) | 36 | 30 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 30 | 66
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: % Time in Stage 2 Sleep at 12 Months, Adjusted for Baseline
Description: Percent of total sleep time spent in Stage 2 sleep at 12 months after adjusting for baseline level of Stage 2 sleep (i.e., baseline value included as a covariate in regression models conducted).
Time Frame: baseline, 12 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Exercise Group | Attention-Control (Health Education) Group
Number analyzed (Participants) | 35 | 30
percentage of sleep time | 53.7 (9.6) | 51.0 (9.8)

2. Secondary Outcome: Sleep Disturbances
Description: Self-reported sleep disturbance subscale on Pittsburgh Sleep Quality Index Subscale consists of 9 items scored on a range of 0 to 3, 0 indicating no disturbance and 3 indicating frequent disturbance.
  All 9 items are summed, and the summary scores is captured by 1 of 4 categories ranging from 0 to 3, with 0 indicating less frequent disturbances and 3 indicating greater frequency of disturbances.
Time Frame: 12 months
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Group | Attention-Control (Health Education) Group
Number analyzed (Participants) | 35 | 30
units on a scale | 1.3 (.47) | 1.6 (.5)

3. Secondary Outcome: Peak Exercise Oxygen Consumption
Description: Peak oxygen consumption measured during symptom limited treadmill exercise stress test
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL of 02 per Kg per minute
Arm/Group | Exercise Group | Attention-Control (Health Education) Group
Number analyzed (Participants) | 35 | 30
mL of 02 per Kg per minute | 24.7 (2.2) | 23.1 (2.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 4-year period
Description: Adverse events were collected by blinded study staff during scheduled clinical measurements (baseline, 6month and 12 month)
Arm/Group | Exercise Group | Attention-Control (Health Education) Group
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/30
Other Adverse Events (participants affected / at risk) | 0/36 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes